CLINICAL TRIAL: NCT03149107
Title: Multimodal Prevention of First Psychotic Episode - a 2x2-Factorial Randomized Trial Investigating the Efficacy of Acetylcysteine and Integrated Preventive Psychological Intervention in Subjects Clinically at High Risk for Psychosis
Brief Title: "Multimodal Prevention of Psychosis - Investigating Efficacy of N-Acetylcysteine and Psychotherapy in CHR-Patients"
Acronym: ESPRIT-B1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment not sufficient
Sponsor: University Hospital, Bonn (Other)
Collaborators: University of Cologne (Other); Central Institute of Mental Health, Mannheim (Other); Ludwig-Maximilians - University of Munich (Other); University Hospital Tuebingen (Other); Heinrich-Heine University, Duesseldorf (Other); Charite University, Berlin, Germany (Other); RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Rene Hurlemann, Professor Dr. Dr. Rene Hurlemann, University Hospital, Bonn
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: University Hospital, Bonn
Record Dates: First submitted 2017-05-08; First posted 2017-05-11 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Prodromal Schizophrenia
Keywords: Prodrome, CHR, Schizophrenia, prevention, N-acetylcysteine
MeSH Terms: conditions — Schizotypal Personality Disorder; Schizophrenia | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IPPI + NAC (Experimental): IPPI (Integrated Preventive Psychological Intervention): 21 sessions, the first 20 sessions are scheduled weekly, the last session two weeks after session 20. Single blinded (statistician & rater).
  N-Acetylcysteine (2000 mg/d, 1000 mg in the morning/evening, oral intake). Will be applied continously over 26 weeks parallel to the psychological intervention. Double-blinded.
  Interventions: Drug: N-Acetylcysteine; Behavioral: IPPI (Integrated Preventive Psychological Intervention)
- PSM + NAC (Experimental): PSM (Psychological stress management): 11 sessions; the first 10 sessions will be offered biweekly, the last one 2 weeks after session 10. Single blinded (statistician & rater).
  N-Acetylcysteine (2000 mg/d, 1000 mg in the morning/evening, oral intake). Will be applied continously over 26 weeks parallel to the psychological intervention. Double-blinded.
  Interventions: Drug: N-Acetylcysteine; Behavioral: PSM (Psychological stress management)
- IPPI + Placebo (Experimental): IPPI (Integrated Preventive Psychological Intervention): 21 sessions, the first 20 sessions are scheduled weekly, the last session two weeks after session 20. Single blinded (statistician & rater).
  Placebo will be applied continously over 26 weeks (oral intake of capsules) parallel to the psychological intervention (IPPI or PSM).
  Interventions: Drug: Placebo; Behavioral: IPPI (Integrated Preventive Psychological Intervention)
- PSM + Placebo (Active Comparator): PSM (Psychological stress management): 11 sessions; the first 10 sessions will be offered biweekly, the last one 2 weeks after session 10. Single blinded (statistician & rater).
  N-Acetylcysteine (2000 mg/d, 1000 mg in the morning/evening, oral intake). Placebo will be applied continously over 26 weeks (oral intake of capsules) parallel to the psychological intervention (IPPI or PSM).
  Interventions: Drug: Placebo; Behavioral: PSM (Psychological stress management)

INTERVENTIONS:
Drug: N-Acetylcysteine — N-Acetylcysteine (2000 mg/d, 1000 mg in the morning/evening, oral intake). Will be applied continously over 26 weeks parallel to the psychological intervention (IPPI or PSM).
  Other Names: NAC
  Arms: IPPI + NAC; PSM + NAC
Drug: Placebo — Will be applied continously over 26 weeks (oral intake of capsules) parallel to the psychological intervention (IPPI or PSM).
  Arms: IPPI + Placebo; PSM + Placebo
Behavioral: IPPI (Integrated Preventive Psychological Intervention) — IPPI (Integrated Preventive Psychological Intervention): 21 sessions, the first 20 sessions are scheduled weekly, the last session two weeks after session 20. Single blinded (statistician & rater)
  Arms: IPPI + NAC; IPPI + Placebo
Behavioral: PSM (Psychological stress management) — PSM (Psychological stress management): 11 sessions; the first 10 sessions will be offered biweekly, the last one 2 weeks after session 10. Single blinded (statistician & rater).
  Arms: PSM + NAC; PSM + Placebo

SUMMARY:
Schizophrenia is a severe mental disorder associated with significant impairments in affective, cognitive and social functioning. Consequently, a special interest in the prevention of schizophrenia and psychotic disorders has emerged. Pharmacological as well as psychological interventions show promising preventive effects. The purpose of this multicentric study is the investigation of possible preventive effects of a treatment combination containing a psychotherapy form and medication (N-Acetylcytein - NAC) in individuals with an enhanced risk for developing schizophrenia. Both treatment forms may reduce the risk in this population due to their specific properties: The psychotherapy can improve social skills, whereas NAC is supposed to develop its protective effects on neuronal level due to its antiinflammatory properties. The investigators will examine the preventive effects by measuring transition rates to psychosis after treatment as well as improvements in social, affective and cognitive functioning.

DETAILED DESCRIPTION:
Psychotic disorders are among the most expensive brain-related disorders in Europe. This is mainly due to their onset early in life and their long-term disabling courses. Current treatments fail to improve most influential factors such as social-cognitive deficits. Prevention is recognized as one of the key strategies to fight these deteriorating outcomes and is expected to significantly reduce both, the societal costs as well as the immense burden for the patients and for their families. Recent meta-analyses indicate promising preventive effects of both pharmacological and cognitive-behavioural interventions. Yet, reported transition rates are still too high. Clinical evidence suggests that disturbances of social functioning predict conversion to psychosis. Neurobiological evidence implicates glutamatergic dysfunction and redox imbalance in the pathophysiology of schizophrenia. The investigators hypothesize that interventions targeting (i) social functioning and (ii) glutamatergic / oxidative pathways already in at-risk states would significantly reduce transition rates. To test these hypotheses, our study is designed as a randomized, placebo-controlled, 18-month trial (six months of intervention plus 12 months of follow-up), involving 200 subjects at-risk for psychosis. Specifically, the investigators will compare the preventive effects of a cognitive-behavioural and social-cognitive intervention to a pharmacological intervention (IPPI) with Acetylcysteine, a drug with a proglutamatergic, neuroprotective and anti-inflammatory profile in a 2x2 factorial design. The results of our planned study are expected to provide new and well tolerated interventions, thus hopefully helping to achieve the major goal of individualized prevention, and, consequently, lower the individual and societal burden of psychosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 40 years;
2. Subjects with the ability to follow study instructions and likely to attend and complete all required visits;
3. Written informed consent of the subject;
4. Subjects are able to speak, write and understand the German language sufficiently well (at the investigators discretion) to complete all required study procedures;

   Specific inclusion criterion:
5. Clinical High Risk Criteria : ESPRIT Ultra-high risk criteria (Attenuated Positive Symptoms and/or Brief Llimited Intermittend Psychotic Symptoms and/or a combination of familial risk or schizotypal disorder with a significant loss of functioning; severity assessed by the Structured Interview for Prodromal Syndromes, SIPS 5.0) and/or The Basic Symptom Criterion 'Cognitive Disturbances, COGDIS' (2/9 cognitive-perceptive basic symptoms; assessed by the Schizophrenia Proneness Instrument - Adult Version, SPI-A)

Exclusion Criteria:

1. Known history of hypersensitivity to the investigational drug or to drugs with a similar chemical structure;
2. Simultaneously participation in another clinical trial involving administration of an investigational medicinal product within 30 days prior to clinical trial beginning. The simultaneous participation in a noninterventional clinical trial is permitted in case the subject is nevertheless able and willing to attend and complete all required visits and in case there are no other contraindications;
3. Subjects with a physical or psychiatric condition which at the investigator's discretion may put the subject at other clinically significant risks than those that are defined as outcome of this study (development of a first psychotic episode, functional deterioration), may confound the trial results, or may interfere with the subject's per protocol participation in this clinical trial;
4. Acute Suicidality;
5. Known substance abuse or dependence according to DSM-IV-TR;
6. Patients with hepatic or renal failure, or with known problems of galactose intolerance, clinically significant lactase deficiency or glucose-galactose malabsorption or histamine-intolerance;
7. Subjects with known asthma bronchiale;
8. Subjects with a history of gastrointestinal ulcer;
9. Intake of antitussives (cough-relieving agents);
10. Intake of nitroglycerin
11. Exclusion criteria regarding special restrictions for females: Current pregnancy or pregnancy planned within 9 months after start of medication or nursing women and
12. Females of childbearing potential, who are not using and not willing to use medically reliable methods of contraception for the entire study duration (such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices) unless they are surgically sterilized / hysterectomized or there are any other criteria considered sufficiently reliable by the investigator in individual cases.

    Indication specific exclusion criteria:
13. Having had a psychotic episode for > 1 week (according to SIPS 5.0);
14. Having symptoms relevant for inclusion potentially arising from a known general medical disorder;
15. Life time antipsychotic medication for more than 30 days (cumulative number of days) at or above minimum dosage of the '1st episode psychosis' range of DGPPN S3 Guidelines (Exception: maximum dosage for aripiprazole 5 mg/d) (Deutsche Gesellschaft für Psychiatrie, Psychotherapie und Nervenheilkunde, 2006);
16. Any intake of antipsychotic medication (i.e., independent of duration of intake) within the past 3 months before psychopathological baseline assessments (including self-ratings and screening assessments) at or above minimum dosage of the '1st episode psychosis' range of DGPPN S3 Guidelines (Exception: maximum dosage for aripiprazole 5 mg/d) (Deutsche Gesellschaft für Psychiatrie, Psychotherapie und Nervenheilkunde, 2006);
17. Any intake of mood stabilizers (lithium, valproate, carbamazepine, oxcabazepine, lamotrigine) > 30 days (cumulative number of days) during the past three months or any intake during the month before psychopathological baseline assessments;
18. Intake of antidepressants during the past 30 days before psychopathological baseline assessments;
19. Intake of benzodiazepines for more than 2 consecutive days during the past 5 days before psychopathological baseline assessments;
20. Psychotherapeutic intervention during the past 30 days before psychopathological baseline assessments;
21. Any past psychotherapeutic treatment targeting specifically psychotic symptoms or its prevention.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Transition to psychosis | I. After intervention phase (26 weeks after trial start) and II. as follow-up (78 weeks after trial start)
  Transition to psychosis within 18 months, defined (according to EPOS1) as the presence of at least one psychotic symptom for at least one week (assessed by the SIPS).
Psychosocial functioning | I. After intervention phase (26 weeks after trial start) and II. as follow-up (78 weeks after trial start)
  Psychosocial functioning assessed by the SOFAS and the FROGS

SECONDARY OUTCOMES:
Symptom remission | I. After intervention phase (26 weeks after trial start) and II. as follow-up (78 weeks after trial start)
  1. Remission of symptomatic clinical high risk (CHR) criteria (APS/BLIPS and/or COGIDS); decrease of positive, negative and disorganization symptoms (assessed by the SIPS, BNSS score); conceptual disorganization and cognitive basic symptoms (COGDIS, SPI-A); as well as at-risk symptoms according to UHR (SPI-A);
Depression remission | I. After intervention phase (26 weeks after trial start) and II. as follow-up (78 weeks after trial start)
  Remission of depressive symptoms (measured by CDSS)
Improvement of social cognition | I. After intervention phase (26 weeks after trial start) and II. as follow-up (78 weeks after trial start)
  Improvement of social cognition (measured by SAT-MC I & II, PoFA)
Assessment of safety and tolerability | I. After intervention phase (26 weeks after trial start) and II. as follow-up (78 weeks after trial start)
  Neurologic and general examination (medical history, weight, - adverse events (assessed by UKU SYMPTOM-LIST), Laboratory assessments

CONTACTS AND LOCATIONS:
Locations (10):
- Germany (10):
  - Zentralinstitut für Gesundheit Mannheim, Mannheim, Baden-Wurttemberg
  - Universitätsklinik Tübingen, Tübingen, Baden-Wurttemberg
  - LMU Klinikum München, München, Bavaria
  - Uniklinik Aachen, Aachen, North Rhine-Westphalia
  - Uniklinikum Bonn, Bonn, North Rhine-Westphalia
  - Uniklinik Köln, Cologne, North Rhine-Westphalia
  - LVR Klinik Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Rheinhessen Fachklinik Alzey, Alzey, Rhineland-Palatinate
  - Charité Berlin, Berlin
  - Berlin Vivantes, Berlin

IPD SHARING:
Plan to Share IPD: Undecided